CLINICAL TRIAL: NCT06083220
Title: School Readiness in Preschool-Aged Children With Cerebral Palsy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Texas Scottish Rite Hospital for Children (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STU-2023-1016
Record Dates: First submitted 2023-10-06; First posted 2023-10-13 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-04

CONDITIONS: Unilateral Cerebral Palsy; School Readiness

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- School Readiness Intervention Program (Experimental): The School Readiness Program is a 64 hour intensive therapy program focused on school readiness skills for young children with unilateral cerebral palsy (UCP). The program will include 64 hours of intervention supporting the development and goal attainment across 5 school readiness domains: (1) health and physical development, (2) emotional well-being and social competence, (3) approaches to learning, (4) communication skills, and (5) cognitive skills and general knowledge.
  Interventions: Behavioral: Smart Start - School Readiness Program

INTERVENTIONS:
Behavioral: Smart Start - School Readiness Program — Participants will complete 64 hours of intervention focused on goal directed school readiness. Each of the five domains will be addressed in each session, and the activities will be tailored to support the individual goals of the participant using a goal-directed training approach. A goal-directed training approach includes the child, caregiver, and researcher collaboratively setting goals that are meaningful to the child and their family. Intervention strategies for goal attainment will include both remediation of skills (i.e. learning to button a button) or the accommodation of skills (i.e. using Velcro instead of a button) depending on the child's goals and current ability. The primary focus of the intervention will be goal attainment related to school readiness.

SUMMARY:
The goal of this feasibility and proof of concept study is to learn about the feasibility, acceptability, and impact of a school readiness program for preschool-aged children with unilateral cerebral palsy. The main question[s] it aims to answer are:

1. Is it feasible to implement an intensive school readiness program for preschool-aged children with UCP?
2. Is the program acceptable to the children and their caregivers?
3. What is the impact of the program on school readiness?

Participants will complete two pre-intervention assessments, participate in an intensive, goal directed, school readiness program, and complete 1 post-intervention assessment.

DETAILED DESCRIPTION:
Introduction and Purpose Cerebral Palsy (CP) is a congenital non-progressive motor disorder caused by a brain lesion that occurs in the early stages of development and persists throughout adulthood. CP is one of the most common disabilities in childhood, with a prevalence of 3.3 per 1,000 children in the United States. It is noted that "children with disabilities have a greater risk of poor or sub-optimal development in early childhood compared to children without disabilities". Due to the nature of CP, the child and their families can experience many limitations in their day-to-day lives and how they participate in their environment. Many of these limitations are brought to light when the child is ready to enter school. It is essential that children with CP and their families understand their child's strengths and areas of need in order to ensure that their child is offered the requisite support services that adequately prepare them for school enrolment. The purpose of this study is to determine if an intensive school readiness program for children with unilateral cerebral palsy (UCP), is feasible and acceptable, and to gain an understanding of the impact of the program on school readiness.

Background "School readiness is a framework for assessing the strengths and vulnerabilities of a child prior to school". Preschool-age children with CP perform significantly lower than their typically developing peers in the areas of mobility, self-care, social function, and communication. Because school readiness is lower in children with disabilities, underachievement and lack of social-emotional skills can further affect how the child develops into adulthood and possibly change the course of their lives. There is very little research regarding school readiness programs specifically for children with cerebral palsy, but other programs that promote school readiness for children on a universal level have shown to be effective.

The school readiness framework can be used to assess a child's strengths and weaknesses in the context of transitioning to entering school. School readiness is the child's ability to participate in 5 major skill areas: (1) health and physical development, (2) emotional well-being and social competence, (3) approaches to learning, (4) communication skills, and (5) cognitive skills and general knowledge. Research indicates children with disabilities encounter challenges in the school setting secondary to poor teacher training, lack of support, decreased social experience, and physical barriers. Understanding the areas that children with CP have deficits in and how we can intervene at an early age can help reduce poor academic performance as the child ages. Studies have shown that providing a school readiness program to any child, typically developing or not, not only increases success in the classroom but can also be an investment in the community's future. School readiness programs can have a positive impact on the community for up to 60 years or more due to increased success of children at an early age carrying on into adulthood. Therefore, there is a need to develop and test a school readiness program that (1) identifies the strengths and areas in need of intervention, (2) educates caregivers on their child's strengths/needs and available resources, and (3) provides intensive therapeutic intervention aimed to address the individual school readiness goals of the child.

Intervention The School Readiness Program is a 64 hour intensive therapy program focused on school readiness skills for young children with unilateral cerebral palsy (UCP). The program will include 64 hours of intervention supporting development and goal attainment across 5 school readiness domains: (1) health and physical development, (2) emotional well-being and social competence, (3) approaches to learning, (4) communication skills, and (5) cognitive skills and general knowledge.

Participants will complete 64 hours of intervention focused on school readiness. Each participant will have an interventionist who is an allied health student with a ratio of 1 child to 1 interventionist or 2 children to 1 interventionist. The interventionists will be trained and overseen by licensed occupational therapists. Each week will have a theme to promote engagement and motivation to participate (i.e. animals, outer space, etc). Each of the five domains will be addressed in each session, and the activities will be tailored to support the individual goals of the participant using a goal-directed training approach. A goal-directed training approach includes the child, caregiver, and researcher collaboratively setting goals that are meaningful to the child and their family. Intervention strategies for goal attainment will include both remediation of skills (i.e. learning to button a button) or the accommodation of skills (i.e. using Velcro instead of a button) depending on the child's goals and current ability. The primary focus of the intervention will be goal attainment related to school readiness. Sessions that are missed due to unexpected or unplanned circumstances (illness, loss of transportation, etc) can be made up via an in-person or virtual session.

Caregivers will be educated on their child's diagnosis, the components of the program, and additional resources that support the child's transition into school. Caregivers will also receive a report including a summary of strengths and areas that are challenging for the child. The goal of the School Readiness program is for children with UCP to increase independence in school readiness activities and to educate the child's caregiver on topics and strategies that will promote a successful transition into school for the child.

ELIGIBILITY:
Inclusion Criteria:

* ages 3 years to 5 years 11 months
* unilateral cerebral palsy
* ability to visually attend to objects
* demonstrates an interest in objects
* attempt to reach for or grasp an item with the impaired upper extremity
* English-speaking participants

Exclusion Criteria:

* uncontrolled epilepsy
* significant visual impairment
* severe behavioral problems
* inability to complete the assessment protocol

Ages: 36 Months to 71 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Estimated)
Dates: Start 2023-12-12 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Canadian Occupational Performance Measure | pre-intervention (within 2 weeks of start of intervention), and within 2 weeks of post-intervention
  The Canadian Occupational Performance Measure is an interview-based assessment of self-perception of performance of everyday living activities (measured on a scale from 1-10 with higher scores representing better performance and higher satisfaction)

SECONDARY OUTCOMES:
Developmental Assessment for Young Children, Second Edition (DAYC-2) | pre-intervention (within 2 weeks of start of intervention), and within 2 weeks of post-intervention
  The Developmental Assessment for Young Children is an interview and observation based norm-referenced developmental assessment (raw scores 0 or 1, converted to standard scores) mean standard score is 100 with a standard deviation of 10. Higher values represent a better outcome.
Assisting Hand Assessment | pre-intervention (within 2 weeks of start of intervention), and within 2 weeks of post-intervention]
  The Assisting Hand Assessment is an observation-based, criterion-referenced assessment that assess bimanual hand function for children with cerebral palsy, aged 18 months-12 years (measured in logits/units on a scale from 0-100). A higher score represents better outcomes.
School Readiness Checklist | pre-intervention (within 2 weeks of start of intervention), and within 2 weeks of post-intervention]
  A parent reported checklist created by the study team to rate the level of independence or mastery their child has with specific tasks within the 5 domains of school readiness (1. health and physical development, 2. emotional well-being and social competence, 3. approaches to learning, 4. communication skills, and 5. cognitive skills and general knowledge). The items on the checklists are commonly recommended by school districts to support success in kindergarten. Items are rated on a scale of 1-4. Higher values represent better outcomes.

OTHER OUTCOMES:
Demographic information | within 2 weeks of start of intervention (pre-intervention)
  Demographic in formation will be collected including: age in years and months, gender, etiology of cerebral palsy, qualitative description of previous exposure to therapy and preschool
Gross Motor Function Classification System (GMFCS) | within 2 weeks of start of intervention (pre-intervention)
  The Gross Motor Function Classification Systems is a 5-level classification system that describes the gross motor function of children and youth with cerebral palsy with 1 being the lowest functioning and 5 being the highest
Manual Ability Classification Scale (MACS) | within 2 weeks of start of intervention (pre-intervention)
  The Manual Ability Classification Scale describes how children with cerebral palsy use their hands during activities of daily living with 1 being the least functional and 5 being the most functional
Communication Function Classification System (CFCS) | within 2 weeks of start of intervention (pre-intervention)
  The Communication Function Classification System is used to classify the everyday communication performance of individuals with cerebral palsy into five levels. Level five has the least ability to effectively send and receive information from another person and level 1 demonstrates effective sending and receiving of information with unfamiliar and familiar people
The Child and Adolescent Scale of Environment | within 2 weeks of start of intervention (pre-intervention)
  The Child and Adolescent Scale of Environment examines the perceived impact (not frequency) of environmental problems (physical, attitudinal, and social) encountered by the child and family. The sum score range is 0-54 with higher scores representing greater extent of environmental problems.
Wechsler Preschool and Primary Scales of Intelligence, 4th Edition (WPPSI-IV) | within 1 month of start of intervention (pre-intervention)
  The WPPSI-IV is a measure of cognitive development including verbal comprehension, visual-spatial, and working memory designed for children ages 2 years 6 months to 7 years 7 months. Standard scores are based on a mean of 100 with a standard deviation of 15. Higher scores represent better outcomes.
Bracken Basic Concept Scale, 4th Edition Receptive (BBCS-4:R) | within 1 month of start of intervention (pre-intervention)
  The BBCS-4:R is a developmental assessment designed to evaluate children's school readiness skills in terms of their understanding of basic concepts that are strongly related to early childhood cognitive and language development as well as early academic achievement including colors, letters, numbers/counting, size/comparison, shapes, and self/social awareness for children ages 3 years to 7 years 11 months. Subtests have scaled scores with a mean of 10 and a standard deviation of 3, composite scores have a mean of 100 with a standard deviation of 15. Higher scores represent better outcomes.
Feasibility and Fidelity Checklist | weekly during the 8 weeks of the intervention
  a form to document intervention session attendance and to document if the key components of the intervention are being implemented on a weekly basis using a yes/no checklist
Participant Engagement and Acceptability Rating Form | weekly during the 8 weeks of intervention
  a form completed by the participant and their caregiver on a weekly basis to rate the acceptability of the intervention sessions and to provide feedback/recommendations for the intervention using likert scaling with 1 being a low rating and 5 being a high rating and open ended qualitative responses

CONTACTS AND LOCATIONS:
Overall Officials: Angela Shierk, PhD, Principal Investigator — Scottish Rite for Children
Locations (1):
- Scottish Rite for Children, Frisco, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Arneson CL, Durkin MS, Benedict RE, Kirby RS, Yeargin-Allsopp M, Van Naarden Braun K, Doernberg NS. Prevalence of cerebral palsy: Autism and Developmental Disabilities Monitoring Network, three sites, United States, 2004. Disabil Health J. 2009 Jan;2(1):45-8. doi: 10.1016/j.dhjo.2008.08.001. PMID 21122742
- [Background] Bourke-Taylor HM, Cotter C, Lalor A, Johnson L. School success and participation for students with cerebral palsy: a qualitative study exploring multiple perspectives. Disabil Rehabil. 2018 Sep;40(18):2163-2171. doi: 10.1080/09638288.2017.1327988. Epub 2017 May 19. PMID 28524702
- [Background] Boyd RN, Novak I, Morgan C, Bora S, Sakzewski L, Ware RS, Comans T, Fahey MC, Whittingham K, Trost S, Pannek K, Pagnozzi A, Mcintyre S, Badawi N, Smithers Sheedy H, Palmer KR, Burgess A, Keramat A, Bell K, Hines A, Benfer K, Gascoigne-Pees L, Leishman S, Oftedal S. School readiness of children at high risk of cerebral palsy randomised to early neuroprotection and neurorehabilitation: protocol for a follow-up study of participants from four randomised clinical trials. BMJ Open. 2023 Feb 27;13(2):e068675. doi: 10.1136/bmjopen-2022-068675. PMID 36849209
- [Background] Gehrmann FE, Coleman A, Weir KA, Ware RS, Boyd RN. School readiness of children with cerebral palsy. Dev Med Child Neurol. 2014 Aug;56(8):786-93. doi: 10.1111/dmcn.12377. Epub 2014 Jan 16. PMID 24433312